CLINICAL TRIAL: NCT04904107
Title: A Multicentre Randomized Controlled Trial to Improve the accUracy of Referrals to the emerGency departmEnt of patieNts With chesT Pain by Using the Modified HEART Score in Emergency Medical Transport (URGENT 2.0)
Brief Title: Improving the Accuracy of Referrals of Patients With Chest Pain
Acronym: URGENT2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VieCuri Medical Centre (Other)
Collaborators: Siemens Healthineers Nederland B.V. (Unknown)
Responsible Party: Principal Investigator, Braim Rahel, Principal investigator, VieCuri Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Study number 2021_002; NL71820.096.19 (Other: Toetsingonline/CCMO)
Record Dates: First submitted 2021-05-11; First posted 2021-05-27 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Chest Pain; Acute Coronary Syndrome; Myocardial Infarction; Myocardial Ischemia; Heart Attack
Keywords: Modified HEART score; Point-of-care testing; Troponin; Siemens Healthineers
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Myocardial Infarction; Myocardial Ischemia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: It concerns an investigator initiated prospective 1:1 randomised clinical trial in chest pain patients in a pre-hospital setting. Patients will be randomised to (A, intervention group) a direct assessment of the modified HEART score (including POC high sensitive troponin measurement) by EMT personnel and refrainment of transport to the cardiac emergency department (ED) in cases of a low score or (B, control group) regular triage and hospital evaluation, taking place at the cardiac ED in the majority of cases.
Who Masked: Care Provider, Investigator
Masking Description: EMT personnel will be blinded for the randomisation sequence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Chest pain patients in the intervention group will be assessed by EMT personnel by performing the modified HEART score (including POC high sensitive troponin-I measurement (POC HS cTnI)) and the referral policy depends on the result.
  * In case of a low modified HEART score (modified HEART 0-3) patients will not be referred to the cardiac ED.
  * Patients with a modified HEART score >3 are directly referred to the cardiac ED after evaluation. These patients will receive standard care.
  Interventions: Diagnostic Test: modified HEART score (including POC hs cTnI analysis)
- Control group (Active Comparator): Chest pain patients in the control group will receive standard triage and standard care according to the local (EMT) protocol.
  Interventions: Other: Standard care and triage according to the local (EMT)protocol.

INTERVENTIONS:
Diagnostic Test: modified HEART score (including POC hs cTnI analysis) — The modified HEART score was developed in 2007 and has been validated to stratify the risk of short-term adverse cardiac events in patients with chest pain at the ED. Negative predictive value (NPV) of the modified HEART score for ACS as well as positive predictive value (PPV) for major adverse cardiac events (MACE) within 6 weeks after presentation is high.
  The modified HEART score is an acronym for history, ECG, age, risk factors and troponin at arrival.The components can be rated 0,1 or 2 points each and result in a total score between 0 and 10.
  Arms: Intervention group
Other: Standard care and triage according to the local (EMT)protocol. — Standard care and triage of chest pain patients according to the local (EMT)protocol.
  Arms: Control group

SUMMARY:
This is a multicenter, prospective, investigator-initiated, randomized controlled trial aiming to reduce the percentage of non-cardiac chest pain (NCCP) patients admitted to the cardiac emergency department (ED) by performing the modified HEART score by emergency medical transport (EMT) personnel.

DETAILED DESCRIPTION:
Patients with acute coronary syndrome (ACS) should be referred to the hospital promptly. However, referring all patients with chest pain is not feasible, as recent studies showed that up to 80% of the patients with acute chest pain do not have ACS.

Bedside point-of-care (POC) high sensitive troponin testing (in fingerprick blood/capillary blood) and the modified HEART score have become available and might play a substantial role in the triage and diagnosis of chest pain patients in a pre-hospital setting by general practitioners (GPs) and EMT personnel in the future. We hypothesize that patients with chest pain can be referred more accurately by using the modified HEART score.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Chest pain or other complaints suspect of ACS for at least 2 hours where the GP or emergency medical personnel are in need of further diagnostics or risk stratification to come to a decision of referral.
* Patients, who have been informed of the nature of the study, agree to its provisions and have provided written informed consent.

Exclusion Criteria:

* Electrocardiographic ST-segment elevation/High suspicion of STE-ACS.
* Suspicion of an acute non-coronary diagnosis e.g. pulmonary embolism, thoracic aortic dissection or other life-threatening disease.
* Patients presenting cardiogenic shock, defined as: systolic blood pressure <90mmHg and heart rate >100 and peripheral oxygen saturation <90% (without oxygen administration)
* Patients presenting with sudden onset heart rhythm disorders and second or third degree atrioventricular block.
* Patients with confirmed ACS, PCI or CABG <30 days prior to inclusion.
* Impaired consciousness defined as an EMV <8.
* Severe shortness of breath.
* Patients with known end-stage renal disease (dialysis and/or MDRD < 30 ml/min).
* Patients with known cognitive impairment.
* Communication issues with patient/language barrier.
* Patients already participating in an interventional cardiology or cardiovascular trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Estimated)
Dates: Start 2021-07-04 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of non-cardiac chest pain (NCCP) patients admitted at the cardiac ED (percentage, %) | 30 days
  Evaluation of the percentage of NCCP patients admitted to the cardiac ED by performing the modified HEART score in comparison to our control group (regular triage and care). We aim to detect a reduction of minimal 10% in unnecessarily referred chest pain patients (NCCP patients) but expect an even higher percentage. A lower percentage of NCCP patients indicates improval of the triage of chest pain patients.
The incidence of MACE (percentage, %) | 30 days, 6 months and 1 year
  The mortality and major adverse cardiovascular events (MACE) i.e. acute myocardial infarction, non-elective percutaneous coronary intervention, coronary artery bypass grafting or all cause death within 30 days, 6 months and 1 year after initial presentation in the intervention group versus control group.
  We aim that the proportion of MACE in the intervention group (modified HEART score) is non-inferior to the control group (regular care and triage). Preliminary results of the second phase of FAMOUS Triage trial showed 15.7% (13.1-18.6) MACE rate.We used the expected incidence of 15.7% as the point estimate (meaning no difference between control and intervention). A higher MACE rate (%) in the intervention group suggests a worst outcome.

SECONDARY OUTCOMES:
The incidence of MACE in subgroups (percentage, %) | 30 days, 6 months and 1 year
  Prespecified subgroup analyses of primary outcomes will be performed for:
  1. Diabetic patients versus non-diabetic patients.
  2. Male versus female patients
  3. Patients referred by GP versus patient referred by triage nurse at GP cooperatives (GPC) versus self referrals.
The incidence of non-cardiac chest pain (NCCP) patients admitted at the cardiac ED in subgroups (percentage, %) | 30 days, 6 months and 1 year
  Prespecified subgroup analyses of primary outcomes will be performed for:
  1. Diabetic patients versus non-diabetic patients.
  2. Male versus female patients
  3. Patients referred by GP versus patient referred by triage nurse at GP cooperatives (GPC) versus self referrals.
Cost-effectiveness analysis | 30 days, 6 months and 1 year
  This economic evaluation investigates the health care costs of full implementation of a prehospital rule- out strategy with the modified HEART score (intervention group) compared with regular care and standard transfer to the hospital to rule out ACS (control group). Health-care costs will be prospectively recorded at baseline and at 30 days follow-up, 6 months and 1 year. This includes health care costs due to readmission, diagnostic testing, revascularization etc. The cost of hospital treatment is determined by the Dutch Diagnose Behandel Combinatie (DBC) hospital reimbursement system and the DBC information system, similar to the international diagnosis related group system.
Assessment of the diagnostic value of the modified HEART score. | 30 days, 6 months and 1 year
  Positive Predictive Value (PPV), sensitivity, specificity and Negative Predictive Value (NPV) of the modified HEART score for ACS will be calculated.
Overview of the actual diagnosis of patients with a low modified HEART score (0-3). | 30 days
  To evaluate the percentage of patients in this specific group with ACS versus no-ACS.
Overview of the actual diagnosis of patients with moderate-high modified HEART score (>3). | 30 days
  To evaluate the percentage of patients in this specific group with ACS versus no-ACS.
Clinical accuracy POC hs cTnI. | 30 days
  Clinical accuracy (Positive Predictive value) of POC hs cTnI assessment versus hs cTnT at the cardiac ED.
Time analysis. | 30 days
  Time elapsed from arrival EMT at patient's home to arrival at ED in intervention group versus control group.

CONTACTS AND LOCATIONS:
Overall Officials: Braim Rahel, Dr., Principal Investigator — Viecuri Medical Centre Northern Limburg; Joan Meeder, Dr., Principal Investigator — Viecuri Medical Centre Northern Limburg; Cees de Vos, Dr., Principal Investigator — Laurentius Hospital Roermond; Arnoud van 't Hof, Prof. dr., Study Director — Zuyderland MC; Robert Willemsen, Dr., Study Director — General practitioner office Nazareth Maastricht
Locations (2):
- Netherlands (2):
  - Laurentius Hospital Roermond, Roermond, Limburg
  - Viecuri Medical Centre Northern Limburg, Venlo, Limburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frenk LDS, Rahel BM, de Vos CB, van Osch FHM, Prestigiacomo FG, Janssen MJW, Willemsen RTA, van 't Hof AW, Meeder JG. Improving the accUracy of Referrals to the emerGency departmEnt of patieNts with chesT pain using the modified HEART score in Emergency Medical Transport (URGENT 2.0): protocol for a multicentre randomised controlled trial. BMJ Open. 2024 Dec 20;14(12):e084139. doi: 10.1136/bmjopen-2024-084139. PMID 39806626